CLINICAL TRIAL: NCT00203502
Title: Primary Systemic Therapy Using Sequential Docetaxel/Cyclophosphamide/Bevacizumab Followed by Doxorubicin in Operable/Locally Advanced Breast Cancer
Brief Title: Primary Systemic Therapy in Operable/Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2004-59
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Operable and Locally advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Cyclophosphamide; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention: Dtx Cyclophosphamide Bev (Experimental): Docetaxel 75m/m2 Cyclophosphamide 500 mg/m2 Bevacizumab 15 mg/kg
  Interventions: Drug: Bevacizumab; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab — IV 15mg/kg 21 days
  Other Names: Avastin
Drug: Cyclophosphamide — 500mg per meter squared, IV every 21 days
  Other Names: Cytoxan
Drug: Docetaxel — 60 mg per meter squared, IV every 21 days
  Other Names: Taxotere; Adriamycin

SUMMARY:
The main purpose of this study is to find out what effects taking the drug bevacizumab together with two chemotherapeutic agents, docetaxel and cyclophosphamide followed by doxorubicin alone before surgery will on breast cancer. Bevacizumab will be given for twelve weeks in combination with chemotherapy then it ill be held during the administration of doxorubicin. Twenty-eight to fifty-six days after undergoing surgery, all patients will receive nine three-weekly infusions of bevacizumab.

DETAILED DESCRIPTION:
Prior to being enrolled in this study, they will undergo an evaluation to determine eligibility. The study doctor will obtain a complete medical history, complete a physical examination including blood pressure and heart rate. The doctor will also obtain a baseline ECG as well as blood tests (approximately two tablespoons of blood). In order to decrease the effects of food, exercise and the sleep/wake cycle variability, all blood samples must be taken between 8AM - 10AM and patients will need to fast (no food or drink) for 10 hours prior to the blood test. Patients will also need to strain from working out prior to the blood test. The study will ask for a list of current medications. Patients will not be eligible if they have a history of or now require long-term anticoagulant (blood thinner) therapy (i.e. Coumadin or anything patients may be taking to prevent blood clots) have an allergy to bevacizumab or any other drugs used in the study.

Many of the following evaluations are commonly done to determine diagnosis and/or stage of breast cancer and may have already had some of all of them done. If the following procedures were not done within three weeks, they will need to be done again prior to receiving any study therapy.

* Diagnosis of breast cancer by fine needle aspiration or core needle biopsy will be required for entry in this study.
* Clip Placement - a clip will be placed in the tumor during the core biopsies as a marker to assist surgeons at the time of surgery.
* Tumor Clip Placements - a caliper is similar to a ruler and is used to measure the tumor from the outside of the body instead of always having to use an ultrasound or MRI.
* Tumor Ultrasound - this is a non-invasive exam that uses sound waves to produce a picture of your tumor.

All study participants will be treated with bevacizumab 15 mg/kg plus docetaxel 75 mg/m2 and cyclophosphamide 500 mg/m2 every three weeks for a total of four treatments. Three weeks after the completion of this part of the treatment patients will start receiving doxorubicin 60 mg/m2 every three weeks for a total of four treatments. All these drugs will be given as intravenous infusion on the first day of each three-week period.

Patients will come in for every three week visits and have a physical exam including blood pressure and heart rate. Medications lists will be taken and any side effects that may have been experienced. Tumor caliper measurements will be done and blood will be drawn at each of these visits.

A mammogram and MUGA scan will be done again just prior to surgery. Patients will undergo tumor surgery approximately six months after treatment. Patients will need to visit the study physician one month after surgery for another physical examination including blood pressure and heart rate, an assessment of any side effects and a list of current medications.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of breast cancer established by biopsy.
* Normal kidney function
* Normal LVEF evaluated by MUGA Scan
* >18 years of age
* Good performance status defined by ECOG scale of 0 or 1
* Consent
* Women of childbearing potential must have a negative pregnancy test.
* Use of effective means of contraception in subjects of child-bearing potential while on treatment and for at least 3 months thereafter.
* Peripheral Neuropathy: must be < grade 1
* Hematologic (minimal values)
* Absolute neutrophil count >1,500/mm3
* Hemoglobin >8.0 g/dl
* Platelet count >100,000/mm3
* Hepatic
* Total bilirubin <ULN
* AST, ALT, Alkaline Phosphatase must be within range

Exclusion Criteria:

* Patients with locally advanced breast cancer with skin ulcerations
* Stage IV breast cancer
* Inflammatory breast cancer
* Allergy to any component of the treatment regimen
* Women who are breast feeding
* Pregnancy or refusal to use effective contraception
* Inability to comply with study and/or follow-up procedures.
* Current, recent, or planned participation in a experimental drug study
* Blood pressure of >150/100 mmHg. Essential hypertension well controlled with anti hypertensives is not an exclusion criterion.
* unstable angina
* New York Heart Association Grade II or greater congestive heart failure
* history of myocardial infarction within 6 months
* history of stroke within 6 months
* Clinical significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastasis
* major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0
* Minor surgical procedure such as fine needle aspirations or core biopsy within 7 days prior to day 0
* Pregnant or lactating
* Urine protein: creatinine ratio >1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Makhoul, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Hsu PC, Kadlubar SA, Siegel ER, Rogers LJ, Todorova VK, Su LJ, Makhoul I. Genome-wide DNA methylation signatures to predict pathologic complete response from combined neoadjuvant chemotherapy with bevacizumab in breast cancer. PLoS One. 2020 Apr 16;15(4):e0230248. doi: 10.1371/journal.pone.0230248. eCollection 2020. PMID 32298288
- [Derived] Makhoul I, Todorova VK, Siegel ER, Erickson SW, Dhakal I, Raj VR, Lee JY, Orloff MS, Griffin RJ, Henry-Tillman RS, Klimberg S, Hutchins LF, Kadlubar SA. Germline Genetic Variants in TEK, ANGPT1, ANGPT2, MMP9, FGF2 and VEGFA Are Associated with Pathologic Complete Response to Bevacizumab in Breast Cancer Patients. PLoS One. 2017 Jan 3;12(1):e0168550. doi: 10.1371/journal.pone.0168550. eCollection 2017. PMID 28045923
- [Derived] Makhoul I, Griffin RJ, Siegel E, Lee J, Dhakal I, Raj V, Jamshidi-Parsian A, Klimberg S, Hutchins LF, Kadlubar S. High-circulating Tie2 Is Associated With Pathologic Complete Response to Chemotherapy and Antiangiogenic Therapy in Breast Cancer. Am J Clin Oncol. 2016 Jun;39(3):248-54. doi: 10.1097/COC.0000000000000046. PMID 24577164
- [Derived] Makhoul I, Klimberg VS, Korourian S, Henry-Tillman RS, Siegel ER, Westbrook KC, Hutchins LF. Combined neoadjuvant chemotherapy with bevacizumab improves pathologic complete response in patients with hormone receptor negative operable or locally advanced breast cancer. Am J Clin Oncol. 2015 Feb;38(1):74-9. doi: 10.1097/COC.0b013e31828940c3. PMID 23563210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients from September 9, 2005 through January 17, 2008. Patients were recruited from hematology/oncology clinic at the Winthrop P. Rockefeller Cancer Institute of the University of Arkansas for Medical Sciences.
Groups:
- Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin: Docetaxel 75mg/m2 + Cyclophosphamide 500 mg/m2
  + Avastin 15 mg/kg
  Q 3 weeks X 4 cycles
  Bevacizumab/Avastin: IV 15mg/kg 21 days
  Cyclophosphamide: 500mg per meter squared, IV every 21 days
  Doxorubicin: 60 mg per meter squared, IV every 21 days
Period: Overall Study
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Started | 40
Completed | 39
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 45 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response.
Description: Pathological complete response was defined as the absence of residual invasive and in situ cancer on hematoxylin and eosin evaluation of the resected breast.
Time Frame: Participants were assessed during surgery, an average of one hour
Measure: Number (90% Confidence Interval); unit: percentage of evaluable patients
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Number analyzed (Participants) | 39
percentage of evaluable patients | 41 [27.7 to 55.4]

2. Secondary Outcome: Number of Participants With Clinical Complete Response in Breast and the Axillary Lymph Nodes After the Completion of Chemotherapy and Bevacizumab.
Description: Clinical complete response was defined using RECIST response categories as the clinical response to chemotherapy
Time Frame: At completion of chemotherapy treatment, an average of one hour
Population: All participants evaluated surgically
Measure: Number (90% Confidence Interval); unit: percentage of pts w/ cCR
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Number analyzed (Participants) | 38
percentage of pts w/ cCR | 53 [39 to 66]

3. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Adverse Events
Description: Percent of participants who had at least one grade 3 or 4 adverse event
Time Frame: After each chemotherapy infusion, approximately one hour
Measure: Number (90% Confidence Interval); unit: percentage of pts w/ grade 3/4 AE
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Number analyzed (Participants) | 39
percentage of pts w/ grade 3/4 AE | 79 [69 to 90]

4. Secondary Outcome: To Measure the Change in Left Ventricular Ejection Fraction (LVEF) From Baseline
Description: Absolute change in LVEF, where LVEF values are measured in percentage units
Time Frame: Immediately before treatment and 1 year after start of treatment
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Number analyzed (Participants) | 34
Percentage of LVEF | -3.5 (7.0)

5. Secondary Outcome: Percentage of Participants With Pathologic Complete Response (pCR) Among Those With Triple Negative Breast Cancer
Description: pCR rate for triple negative patients--percent
Time Frame: at surgery, one day
Population: Patients with triple negative breast cancer
Measure: Number (90% Confidence Interval); unit: % pCR among triple negative pts
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Number analyzed (Participants) | 14
% pCR among triple negative pts | 57 [35 to 79]

ADVERSE EVENTS:
Description: If a subject experienced more than 1 of a given AE, the subject is only counted once for that AE. If a subject experienced more than one AE is a system organ class, the subject is only counted once in that system organ class.
Arm/Group | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin
Serious Adverse Events (participants affected / at risk) | 39/39
Other Adverse Events (participants affected / at risk) | 19/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin (N=39)
infection (Infections and infestations) | 3 (3)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Fatigue (General disorders) | 4 (8)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Drug:Docetaxel + Cyclophosphamide + Avastin (N=39)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (19)
Constipation (Gastrointestinal disorders) | 19 (19)
Fatigue (General disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes